CLINICAL TRIAL: NCT00437450
Title: Treatment of the Anemia of Myelodysplastic Syndromes by the Association of Epoetin Beta and All Trans Retinoic Acid
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Groupe Francophone des Myelodysplasies (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 040759
Record Dates: First submitted 2007-02-19; First posted 2007-02-21 (Estimated); Last update posted 2009-11-18 (Estimated); Status verified 2007-02

CONDITIONS: Anemia in Myelodysplastic Syndromes
Keywords: Anemia; myelodysplastic syndromes; Low risk; Bone Marrow diseases
MeSH Terms: conditions — Anemia; Myelodysplastic Syndromes; Bone Marrow Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Epoetin/Atra

SUMMARY:
The purpose of this study is

* To evaluate the efficacy of association of Erythropoetin (Neorecormon) and ATRA in patients with low risk myelodysplastic syndromes
* To evaluate the tolerance of this treatment

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years with RA, RARS, RAEB (blasts <10%)
* Hb< 10g/dl > of 2 months or transfused since less 2 months
* Hb<12g/dl > of 2 months and thrombocytopenia defined by platelets < 50 000/mm3, or neutropenia<10 000mm3
* For women of child bearing age, necessity of contraception during all the duration of the study

Exclusion Criteria:

* Patient with lung disease, cardiac, neurological, gastro-intestinal or genito - urinary disorders not connected to genito -urinary not connected to myelodysplasia
* Patient having received intensive chemotherapy in the 3 months before inclusion in the protocol
* RAEBt
* RAEB >10% blasts
* Treatment with rHu-Epo, darbepoetin ou rHu-GCSF , 2 months before inclusion
* Patient presenting an iron , B12 vitamin or folic acid uncorrected deficit
* CMML
* Uncontrolled systemic hypertension
* creatinine clearance < 300 µM/L
* Pregnant patient or in period of lactation
* Life expectancy < 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99
Dates: Start 2004-10; Study Completion 2005-09

PRIMARY OUTCOMES:
To evaluate the efficacy of association of Erythropoetin and ATRA in patients with low risk myelodysplastic syndromes

SECONDARY OUTCOMES:
To evaluate the tolerance of this treatment

CONTACTS AND LOCATIONS:
Overall Officials: Lionel ADES, MD, Principal Investigator — Groupe Francophone des Myelodysplasies
Locations (24):
- France (24):
  - CHU d'Amiens, Amiens
  - CHU d'Angers, Angers
  - CHU d'Avignon, Avignon
  - CH de la cote Basque, Bayonne
  - Hopital Avicenne, Bobigny
  - CHU de Caen, Caen
  - Hopital Percy, Clamart
  - CHU Dijon, Dijon
  - CHU Albert Michallon, Grenoble
  - CHRU Limoges, Limoges
  - CHU Edouard Herriot, Lyon
  - Institut Paoli Calmette, Marseille
  - CHU Archet, Nice
  - Hopital Necker, Paris
  - Hopital Saint Antoine, Paris
  - HOPITAL Cochin, Paris
  - Hopital Hotel Dieu, Paris
  - CH de Cournouaille, Quimper
  - CHU Robert Debre, Reims
  - Hopital Henri Becquerel, Rouen
  - Hopital Hautepierre, Strasbourg
  - Chu Purpan, Toulouse
  - CHU Bretoneau, Tours
  - CHU Brabois, Vandœuvre-lès-Nancy